CLINICAL TRIAL: NCT03253198
Title: Preoperative Interscalene Nerve Block Plus Postoperative Local Intra-operative Analgesic Injection vs Preoperative Interscalene Nerve Block Plus Postoperative Saline Injection in Patients Undergoing Shoulder Arthroplasty: a Randomized Trial
Brief Title: Prospective RCT Comparing Perioperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017SNam
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Arthroplasty Shoulder
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preoperative block plus saline (Active Comparator): Preoperative interscalene brachial plexus single-shot block using 25ml of 0.5% Ropivicaine plus postoperative 40cc local infiltration of saline
  Interventions: Drug: Saline
- Preoperative block plus Bupivacaine extended-release liposome (Active Comparator): Interscalene brachial plexus single shot block preoperatively (25 ml of 0.5% ropivicaine) + Postoperative Infiltration of local anesthetic/analgesic (20 cc Bupivacaine extended-release liposome injection (Exparel) + Diluted in 20cc of Saline into the capsule, subscapularis, deltoid, pectoralis major and subcutaneous tissues)
  Interventions: Drug: Bupivacaine liposome

INTERVENTIONS:
Drug: Saline — A preoperative interscalene brachial plexus single-shot block using 25 ml of 0.5% Ropivicaine plus saline injection postoperative
  Arms: Preoperative block plus saline
Drug: Bupivacaine liposome — an interscalene brachial plexus single shot block preoperatively (25 ml of 0.5% ropivicaine) + Postoperative Infiltration of local anesthetic/analgesic (20 cc Bupivacaine extended-release liposome injection (Exparel) + Diluted in 20cc of Saline into the capsule, subscapularis, deltoid, pectoralis major and subcutaneous tissues)
  Arms: Preoperative block plus Bupivacaine extended-release liposome

SUMMARY:
This study is a non-blinded randomized controlled trial comparing the use of a preoperative "mini" block plus postoperative local infiltration of Exparel (liposomal form of bupivacaine) versus a partial single shot nerve block in subjects undergoing primary reverse or total shoulder arthroplasty to see which is more effective in controlling surgery related pain. To do so, we will utilize the Visual Analog Scale (VAS) to measure pain intensity. Opioid consumption will be recorded on a Pain Monitoring Sheet.

ELIGIBILITY:
Inclusion Criteria:

* All individuals undergoing primary reverse and total shoulder arthroplasty by the shoulder service at Thomas Jefferson University Hospital, Methodist Hospital or Rothman Specialty Hospital.

Exclusion Criteria:

* Psychiatric illness as defined by co-morbid diagnosis of bipolar disorder or schizophrenia
* Revision arthroplasty or arthroplasty for fracture
* Unable/unwilling to consent for enrollment
* Unable to complete postoperative pain survey
* Known adverse drug reaction or allergy to the medications used
* Chronic pain syndromes (including reflex sympathetic dystrophy, fibromyalgia, chronic diffuse musculoskeletal pain)
* Patients taking long acting opioid pain medications (including extended release opioid pain medications and methadone)
* Patients under the age of 18 years
* Patients with history of hepatic disease
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
morphine and morphine equivalent consumption | 24 hours post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Surena Namdari, MD, Principal Investigator — Rothman Institute
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No